CLINICAL TRIAL: NCT04389593
Title: Comparative and Additive Diagnostic Performance of Magnetic Resonance Elastography (MRE) and Corrected-T1 (cT1) for Fibrosis and Inflammation in Nonalcoholic Steatohepatitis (NASH) Using Histology As Reference
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Claude Sirlin, Professor, University of California, San Diego
Other Study IDs: 181449
Record Dates: First submitted 2020-02-26; First posted 2020-05-15 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-08

CONDITIONS: Nonalcoholic Fatty Liver; Nonalcoholic Steatohepatitis; Liver Fibroses; Liver Inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Cirrhosis; Hepatitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Single arm: This is a single arm study in which all participants have one MRI

SUMMARY:
This pilot study will evaluate conventional and investigational MR imaging and spectroscopic sequences and collect data to help plan more definitive future studies.

DETAILED DESCRIPTION:
This prospective pilot study evaluates the comparative and additive diagnostic performance of Magnetic Resonance Elastography (MRE) and corrected-T1 (cT1) for the detection and staging of fibrosis and inflammation in Nonalcoholic Steatohepatitis (NASH), using histology as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects of any gender and any ethnic group with known or suspected NASH
* Subject is willing and able to complete required research procedures (screening/enrollment, clinical evaluation, safety procedures, and research MRI exam), and is willing to allow the study team to review clinical data including but not limited to other clinical radiology reports and images and clinical or research biopsy results
* Subject has been fully informed and has personally signed and dated the written Informed Consent and Health Insurance Portability and Accountability Act (HIPAA) documents
* Subject has had or is expected to have a clinical or research biopsy within 150 days of the MR exam

Exclusion Criteria:

* VA subject
* < 18 years of age
* Subject does not have a physician and does not wish to be contacted about possible incidental findings
* MRI contraindication(s)
* Subject knows that she is pregnant or states she is trying to become pregnant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with known or suspected NASH
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
Accuracy of MRE and c-T1 to assess disease progress | up to one year
  The positive predictive value of quantitative imaging will be compared to histology for the assessment of NASH.

CONTACTS AND LOCATIONS:
Overall Officials: Claude B Sirlin, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No